CLINICAL TRIAL: NCT02838251
Title: Effects of Compression in Mixed Ulcers
Acronym: ULCEREMIXTE
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ULCERE MIXTE
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Ulcer
MeSH Terms: conditions — Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention

SUMMARY:
About 15% to 30% of patients with venous leg ulcers have a peripheral arterial disease (PAD) associated. The compression band is still a controversial issue in this context. It allows the reduction of venous hypertension and edema, but it could potentially degrade the arterial infusion of high levels of compression. The French High Authority for Health (HAS) defines mixed ulcers by IPS between 0.5 and 0.9. Investigators distinguish mixed ulcers blood predominance for IPS between 0.5 and 0.7; and mixed ulcers predominantly venous blood with moderate involvement for IPS values between 0.7 and 0.9.

Several studies have shown that IPS> 0.8 allowed a high compression, between 30 and 40 mmHg. In the case of mixed ulcers with IPS between 0.6 and 0.8, the HAS recommends using a lighter compression, bit by elastic bands (exercising low power compression at rest) under medical supervision, informing the patient to remove the bandage if pain or aggravation. It is therefore necessary to adapt the compression therapy in case of venous ulcers associated with arterial disease by providing a lower compression 30 mmHg short stretch. For HAS, IPS <0.6 against indicates compression.

A recent study showed that compression bit elastic bands could not only improve venous return, but it would also increase the distal arterial flow in a patient population with mixed ulcers. In this study, 25 patients had between IPS 0.5 and 0.8; or for certain patients below the threshold of 0.6 indicates that against a compression according to HAS. To our knowledge this is the only study that has examined the effect of compression on blood perfusion.

DETAILED DESCRIPTION:
Objectives:

* Principal: Study the distal arterial infusion in a patient population with mixed ulcers under compression leg with little elastic bands
* Secondary: To evaluate the safety of the little compression elastic band in a mixed population of patients with leg ulcers

Methodology :

* Study non-interventional prospective single-center that evaluates professional practice from 25 patients with mixed leg ulcers and followed in the vascular medicine department of St. Joseph Hospital Group Paris.
* Applying a bit compression elastic bandages to a pressure level between 30 and 40mmHg.
* Anonymous data reports on the grid standardized collection, by a numbering system from 1 to 30 and then captured on a computer file

  * Age, risk factors and cardiovascular history of the patients,
  * Age, ulcer description
  * Palpation of pulse
  * morphological vascular profile of patients with arterial and venous Doppler dating less than a year,
  * Series following data before installation, 10 minutes after application and 24 hours after installation of the inelastic compression:

    o Evaluation of tolerance:
  * measurement of pain numeric scale (NS)
  * description of the skin condition of the leg by a dermatologist, seeking signs of suffering skin after application of compression: possible appearance of erythema, cyanosis, purpura. A search particularly in areas of bony prominences and the banks of the ulcer.

    o distal arterial pressures of the compression carrier leg:
  * IPS (systolic pressure index): ankle and arm pressures will be measured with a cuff and a continuous Doppler. GPI is calculated by dividing the lowest pressure at the ankle (at the dorsalis pedis or posterior tibial artery) by the humeral pressure.
  * Transcutaneous Oxygen Pressure (TcPO2) o Measuring pressure exerted by low elastic bandages by Kikuhime® system.

In case of bad tolerance of compression at any time after installation, the compression will be removed and the study stopped for the patient in question. Poor tolerance is defined by an increase in pain than or equal to 2 points on the digital scale.

expected benefits for patients:

* Demonstration of good tolerance, defined as no worsening of the skin condition and the lack of increase in pain associated with inelastic compression.
* Demonstration of no worsening of arterial infusion by inelastic compression.
* Evidence of improved distal arterial hemodynamics (increased IPS and tcpO2) with a little elastic compression, which validate the results of the only study ever conducted on the subject.

ELIGIBILITY:
The mixed origin of the ulcer is defined by a venous disease (reflux in the superficial veins and / or deep) and a moderate arterial disease, defined by:

Inclusion Criteria:

* A IPS 0.5 and 0.9, with a systolic pressure at the ankle> 70 mmHg
* A big toe pressure index (IPGO) <0.7, with a systolic pressure of the big toe (PGO)> 50 mmHg

Exclusion Criteria:

* Topics aged under 18,
* A normal IPS that is to say between 0.9 and 1.3, a critical ischemia (defined as ankle pressure <70 mmHg and / or systolic pressure of the big toe <50 mmHg)
* Presence of peripheral neuropathy,
* Presence of heart failure,
* Refusal to participate in the study or to sign the consent,
* Impaired cognitive function not to participate in a clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects older than 18 years, suffering from an ulcer of mixed origin leg, and followed in the vascular medicine department of St. Joseph Hospital Group Paris.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Assessment of change of pain numeric scale | Day 1, just before the exam, 10minutes after the exam and 24 hours after the exam

SECONDARY OUTCOMES:
Assessment of change of distal arterial pressures of the compression carrier leg | Day 1, just before the exam, 10minutes after the exam and 24 hours after the exam
Assessment of change of IPS (systolic pressure index) ankle pressures | Day 1, just before the exam, 10minutes after the exam and 24 hours after the exam
Assessment of change of pressure exerted by low elastic bandage | Day 1, just before the exam, 10minutes after the exam and 24 hours after the exam
  Measuring pressure exerted by low elastic bandages by Kikuhime® system.
Assessment of IPS (systolic pressure index) arm pressures | Day 1, just before the exam, 10minutes after the exam and 24 hours after the exam

CONTACTS AND LOCATIONS:
Overall Officials: STANSAL Audrey, MD, Principal Investigator — Groupe Hospitalier Paris Saint-Joseph (FRANCE)
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided